CLINICAL TRIAL: NCT02078856
Title: A Phase II, Placebo-controlled, Multi-centre, Dose-finding Efficacy and Safety Study of a Range of Doses of A3384 in Patients With Bile Acid Malabsorption (BAM)/Bile Acid Diarrhoea (BAD)
Brief Title: Double-blind, Randomised Study of A3384 in BAM/BAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3384-001
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Bile Acid Malabsorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A3384 Low dose (Experimental): Administered twice daily for the duration of the study
  Interventions: Drug: A3384
- A3384 High dose (Experimental): Administered twice daily for the duration of the study
  Interventions: Drug: A3384
- Placebo (Placebo Comparator): Administered twice daily for the duration of the study
  Interventions: Drug: A3384

INTERVENTIONS:
Drug: A3384

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of A3384 administered to patients with Bile Acid Malabsorption (BAM)/Bile Acid Diarrhoea (BAD).

ELIGIBILITY:
Inclusion Criteria:

* Patient meets protocol specified criteria for Bile Acid Malabsorption/Bile Acid Diarrhoea
* Patient has successfully completed study requirements with no clinically relevant findings for physical exam, ECG, laboratory tests as applicable

Exclusion Criteria:

* Medical history or medical condition that would not make the patient a good candidate for the study or limit the patient´s ability to complete the study
* Patient needs medications prohibited as specified in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective of this study is to demonstrate the efficacy of different daily doses of A3384 as determined by the # of bowel movements (BMs). | 2 weeks

SECONDARY OUTCOMES:
Secondary efficacy objectives of this study are to demonstrate the efficacy of different daily doses on other BM parameters and BAM/BAD symptoms | Baseline and 2 weeks
  Change from Baseline in average severity of diarrhoea during the second treatment week (last 7 days of reporting).
  * Change from Baseline in average severity of abdominal discomfort during the second treatment week (last 7 days of reporting).
  * Change from Baseline in average severity of abdominal bloating during the second treatment week (last 7 days of reporting).
  * Change from Baseline in average BSFS during the second treatment week (last 7 days of reporting)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- Sweden (2):
  - Sahlgrenska Academy, Gothenburg
  - Kärnsjukhuset, Skövde
- Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants. Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/